CLINICAL TRIAL: NCT00708201
Title: A Phase 4, Multicenter, Double-Blind, Placebo-Controlled, Parallel Study of Alvimopan for the Management of Postoperative Ileus in Subjects Undergoing Radical Cystectomy.
Brief Title: A Study of Alvimopan for the Management of Postoperative Ileus in Participants Undergoing Radical Cystectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3753-002; 14CL403 (Other: Cubist Study Number)
Record Dates: First submitted 2008-06-27; First posted 2008-07-02 (Estimated); Results first posted 2015-07-02 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Postoperative Ileus
Keywords: ileus; POI
MeSH Terms: conditions — Ileus | interventions — alvimopan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alvimopan (Experimental): 12 milligrams (mg)
  Alvimopan, 12mg, capsule. Administered orally. One 30 minutes to 5 hours before the scheduled start of surgery on Day 0, and twice daily beginning on Postoperative Day 1 (POD 1) until hospital discharge or for a maximum of 7 days (up to 15 doses) of postoperative treatment
  Interventions: Drug: Alvimopan
- Placebo (Placebo Comparator): 300 mg polyethylene glycol in a capsule
  Administered orally at least 30 minutes and no later than 5 hours before the scheduled start of surgery on Day 0. On Day 1, a single dose of placebo was given twice a day for a maximum of 7 days in hospital after surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alvimopan
  Other Names: ADL2698; Entereg
  Arms: Alvimopan
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study is being conducted to determine whether alvimopan can accelerate recovery of gastrointestinal function following radical cystectomy when compared with a placebo. Secondary objectives of the study are:

* to evaluate the effect of alvimopan on hospital length of stay
* to evaluate the effect of alvimopan on prespecified postoperative ileus (POI)-related morbidities
* to evaluate the overall and cardiovascular safety of alvimopan

ELIGIBILITY:
Inclusion Criteria:

* are either Male or Female at least 18 years of age
* are scheduled for radical cystectomy
* are scheduled to receive postoperative pain management with intravenous participant-controlled opioid analgesics

Exclusion Criteria:

* are scheduled for a partial cystectomy
* have taken more than 3 doses of opioids (oral or parenteral) within 7 days before the day of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2009-03; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Techner, DPM, Study Director — Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)
Locations (20):
- United States (20):
  - Saddleback Memorial Medical Center, Laguna Hills, California
  - University of Colorado Hospital, Aurora, Colorado
  - University of Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - The University of Chicago Medical Center, Chicago, Illinois
  - University of Chicago, Section of Urology MC6038, Chicago, Illinois
  - Indiana University Hospital, Indianapolis, Indiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Michigan Health System, Ann Arbor, Michigan
  - University of Minnesota Hospital, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - CRC of Jackson, Jackson, Mississippi
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Bend Memorial Clinic, Bend, Oregon
  - Oregon Health and Science University Knight Cancer Institute, Portland, Oregon
  - Vanderbilt University Medical Center, Department of Urology Surgery, Nashville, Tennessee
  - The Methodist Hospital, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Lee CT, Chang SS, Kamat AM, Amiel G, Beard TL, Fergany A, Karnes RJ, Kurz A, Menon V, Sexton WJ, Slaton JW, Svatek RS, Wilson SS, Techner L, Bihrle R, Steinberg GD, Koch M. Alvimopan accelerates gastrointestinal recovery after radical cystectomy: a multicenter randomized placebo-controlled trial. Eur Urol. 2014 Aug;66(2):265-72. doi: 10.1016/j.eururo.2014.02.036. Epub 2014 Feb 26. PMID 24630419

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: A single dose of placebo was administered orally at least 30 minutes and no later than 5 hours before the scheduled start of surgery on Day 0. On Day 1, a single dose of placebo was given twice a day for a maximum of 7 days in hospital after surgery.
- Alvimopan 12 mg: A single dose of alvimopan 12 milligrams (mg) was administered orally at least 30 minutes and no later than 5 hours before the scheduled start of surgery on Day 0. On Day 1, a single dose of alvimopan 12 mg was given twice a day for a maximum of 7 days in hospital after surgery.
Period: Overall Study
Arm/Group | Placebo | Alvimopan 12 mg
Started | 137 | 143
Received at Least 1 Dose of Study Drug | 130 | 137
Completed | 130 | 137
Not Completed | 7 | 6
Not completed — Adverse Event | 4 | 4
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: All study participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Alvimopan 12 mg | Total
Number analyzed (Participants) | 137 | 143 | 280
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.9 (9.84) | 66.3 (10.93) | 65.1 (10.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 30 | 57
  Male | 110 | 113 | 223
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 134 | 142 | 276
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 6 | 4 | 10
  White | 131 | 138 | 269
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Time to Achieve GI2 Analyzed by Kaplan-Meier (KM) Estimates and Cox Proportional Hazards (PH) Model
Description: Time to achieve recovery of gastrointestinal (GI) function as measured by a composite endpoint of both upper GI recovery (toleration of solid food) and lower GI recovery (first bowel movement [BM]) using KM Estimates and Cox PH Model. This endpoint was referred to as GI2. GI2 was calculated as GI2 = maximum (max) (solids, BM). The KM estimate reported below is biased because of the censoring of the last observation.
  Censoring Rules for Study Participants who:
  Completed: the censored time for the event was determined as: censored time = minimum [maximum (time of/to last GI assessment, time of/to hospital discharge order written), study duration].
  Discontinued: censored time = maximum (time of/to last GI assessment, time of/to discontinuation)
Time Frame: From day of surgery (Day 0) up to 10 days in hospital
Population: All participants who received at least 1 dose of study medication, who had at least 1 postdose GI assessment, who had the protocol-specified surgery, and had evaluable time to achieve G12 data. 39 participants in the Placebo group and 17 participants in the Alvimopan group were censored.
Measure: Mean (Standard Error); unit: Hours
Arm/Group | Placebo | Alvimopan 12 mg
Number analyzed (Participants) | 134 | 143
Hours | 164.2 (5.56) | 132.7 (4.30)
Statistical Analysis 1: Comparison: Placebo vs Alvimopan 12 mg; Test type: Superiority or Other; p < 0.0001, Wald's Chi-Square; Hazard Ratio (HR) = 1.773, 95% CI 2-sided [1.359 to 2.311]

2. Secondary Outcome: Mean Time to Ready for Discharge From Hospital Analyzed by KM Estimates and Cox PH Model
Description: The endpoint of "time to ready for discharge" was based solely on the recovery of GI function as determined by the surgeon. The KM estimate reported below is biased because of the censoring of the last observation.
  Censoring Rules for Study Participants who:
  Completed: the censored time for the event was determined as: censored time = minimum [maximum (time of/to last GI assessment, time of/to hospital discharge order written), study duration].
  Discontinued: censored time = maximum (time of/to last GI assessment, time of/to discontinuation)
Time Frame: Day of surgery (Day 0) up to 10 days in hospital
Population: All participants who received at least 1 dose of study medication, who had at least 1 postdose GI assessment, who had the protocol-specified surgery, and had evaluable ready to discharge data. 21 participants in the Placebo group and 12 participants in the Alvimopan group were censored.
Measure: Mean (Standard Error); unit: Hours
Arm/Group | Placebo | Alvimopan 12 mg
Number analyzed (Participants) | 134 | 143
Hours | 154.7 (5.28) | 130.0 (4.15)
Statistical Analysis 1: Comparison: Placebo vs Alvimopan 12 mg; Test type: Superiority or Other; p < 0.001, Log Rank; Mean Difference (Final Values) = -24.7, 95% CI 2-sided [-37.8 to -11.5]

3. Secondary Outcome: Mean Time to Discharge Order Written (DOW) Using KM Estimates
Description: The KM estimate reported below is biased because of the censoring of the last observation.
  Censoring Rules for Study Participants who:
  Completed: the censored time for the event was determined as: censored time = minimum [maximum (time of/to last GI assessment, time of/to hospital discharge order written), study duration].
  Discontinued: censored time = maximum (time of/to last GI assessment, time of/to discontinuation)
Time Frame: Day of surgery (Day 0) up to 10 days in hospital
Population: All participants who received at least 1 dose of study medication, who had at least 1 postdose GI assessment, who had the protocol-specified surgery, and had evaluable time to DOW data. 36 participants in the Placebo group and 15 participants in the Alvimopan group were censored.
Measure: Mean (Standard Error); unit: Hours
Arm/Group | Placebo | Alvimopan 12 mg
Number analyzed (Participants) | 134 | 143
Hours | 188.4 (5.11) | 166.0 (3.89)
Statistical Analysis 1: Comparison: Placebo vs Alvimopan 12 mg; Test type: Superiority or Other; p < 0.001, Log Rank; Mean Difference (Final Values) = -22.4, 95% CI 2-sided [-35.0 to -9.9]

4. Secondary Outcome: Postoperative Length of Stay (LOS)
Description: The postoperative LOS was determined by the difference between the date of hospital DOW and the date of surgery; that is, the postoperative LOS for a participant was calculated as follows: (date of DOW) - (date of surgery).
Time Frame: Day of surgery (Day 0) to the day of hospital DOW
Population: All participants who received at least 1 dose of study medication, who had at least 1 postdose GI assessment, who had the protocol-specified surgery, and had evaluable postoperative LOS data.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | Alvimopan 12 mg
Number analyzed (Participants) | 134 | 143
Days | 10.07 (8.23) | 7.44 (3.05)
Statistical Analysis 1: Comparison: Placebo vs Alvimopan 12 mg; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Percentage of Participants Considered Postoperative LOS Responders
Description: A participant was considered a postoperative LOS responder if the postoperative LOS was less than or equal to 7 days. The postoperative LOS for a participant was calculated as follows: (date of DOW) - (date of surgery). Participants with missing data were considered nonresponders.
Time Frame: Day of surgery (Day 0) up to 7 days after surgery
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alvimopan 12 mg
Number analyzed (Participants) | 134 | 143
percentage of participants | 48.5 | 67.1
Statistical Analysis 1: Comparison: Placebo vs Alvimopan 12 mg; Test type: Superiority or Other; p < 0.01, Fisher Exact; Relative Risk = 1.38, 95% CI 2-sided [1.12 to 1.71] — This is the relative risk for being a responder (alvimopan/placebo)

6. Secondary Outcome: Percentage of Participants With Postoperative Morbidity (POM)
Description: POM was defined as the need for postoperative nasogastric (NG) tube insertion, hospital stay prolonged because of postoperative ileus (POI) (as determined by the investigator), or readmission (readmiss) to the hospital (hosp) for POI within 7 days (d) after discharge.
Time Frame: During hospitalization or within 7 days after discharge
Population: All participants who received at least 1 dose of study medication, who had at least 1 postdose GI assessment, who had the protocol-specified surgery, and had evaluable POM data.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alvimopan 12 mg
Number analyzed (Participants) | 134 | 143
percentage of participants
  Overall POM (n=134, 143) | 29.1 | 8.4
  Postoperative NG tube insertion (n=134, 143) | 24.6 | 7.7
  Prolonged hospital stay due to POI (n=133, 143) | 21.8 | 3.5
  POI rslt in readmiss to hosp in ≤7days(n=134,143) | 0.8 | 0.7
Statistical Analysis 1: Comparison: Placebo vs Alvimopan 12 mg; Statistical analysis for overall POM is presented; Test type: Superiority or Other; p < 0.001, Fisher Exact; Percent difference = -20.71 — Percent difference = alvimopan - placebo

7. Secondary Outcome: Percentage of Participants Considered G12 Responders at 5 Cutoff Time Points
Description: Time to achieve recovery of GI function was measured by a composite endpoint of time to first BM and time to tolerate first solid food (solids). This endpoint was referred to as GI2, and GI2 was calculated as follows: GI2 = max (solids, BM). GI2 responders were defined as those participants who met all the following criteria: achieved GI2 by the cutoff point, did not have hospital stay prolonged because of POI, and did not have readmission for POI within 7 days of actual hospital discharge. Postsurgery Days (PSD) were measured in 24 hour increments after surgery.
Time Frame: Day of surgery (Day 0) through PSD 3, PSD 4, PSD 5, PSD 6, and PSD 7
Population: All participants who received at least 1 dose of study medication, who had at least 1 postdose GI assessment, who had the protocol-specified surgery, and had evaluable time to achieve G12 data.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alvimopan 12 mg
Number analyzed (Participants) | 134 | 143
percentage of participants
  PSD 3 | 9.7 | 25.2
  PSD 4 | 27.6 | 53.8
  PSD 5 | 42.5 | 75.5
  PSD 6 | 53.0 | 79.7
  PSD 7 | 57.5 | 84.6
Statistical Analysis 1: Comparison: Placebo vs Alvimopan 12 mg; Statistical analysis for day of surgery (Day 0) through PSD 7 is presented; Test type: Superiority or Other; p < 0.0001, Fisher Exact; Percent difference = 27.05 — Percent difference = alvimopan - placebo

8. Secondary Outcome: Percentage of Participants Considered DOW Responders at 5 Cutoff Time Points
Description: DOW responders were defined as those participants who met all the following criteria: achieved DOW by the cutoff point, did not have hospital stay prolonged because of POI, and did not have readmission for POI within 7 days of actual hospital discharge. PSD were measured in 24 hour increments after surgery.
Time Frame: Day of surgery (Day 0) through PSD 3, PSD 4, PSD 5, PSD 6, and PSD 7
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alvimopan 12 mg
Number analyzed (Participants) | 134 | 143
percentage of participants
  PSD 3 | 0.7 | 2.8
  PSD 4 | 17.9 | 14
  PSD 5 | 32.1 | 39.9
  PSD 6 | 47.8 | 62.2
  PSD 7 | 55.2 | 80.4
Statistical Analysis 1: Comparison: Placebo vs Alvimopan 12 mg; Statistical analysis for day of surgery (Day 0) through PSD 7 is presented; Test type: Superiority or Other; p < 0.0001, Fisher Exact; Percent difference = 25.20 — Percent difference = alvimopan - placebo

9. Secondary Outcome: Percentage of Participants With Blinded Adjudicated Cardiovascular (CV) Events
Description: CV events of interest included congestive heart failure, CV death, cerebrovascular accident, myocardial infarction, serious arrhythmia, and unstable angina. CV events were adjudicated by a blinded external committee.
Time Frame: Baseline to 30 days post discharge
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alvimopan 12 mg
Number analyzed (Participants) | 137 | 143
percentage of participants
  Overall CV events of interest | 15.3 | 8.4
  Congestive heart failure | 2.9 | 0.0
  CV death | 2.9 | 0.7
  Cerebrovascular accident | 0.7 | 0.7
  Myocardial infarction | 7.3 | 2.8
  Serious arrhythmia | 5.1 | 5.6
  Unstable angina | 0.7 | 0.7
Statistical Analysis 1: Comparison: Placebo vs Alvimopan 12 mg; Test type: Superiority or Other; p = 0.0946, Fisher Exact; Percent difference = -6.94, 95% CI 2-sided [-14.5 to 0.62] — Percent difference = alvimopan - placebo

ADVERSE EVENTS:
Arm/Group | Placebo | Alvimopan 12 mg
Serious Adverse Events (participants affected / at risk) | 67/137 | 51/143
Other Adverse Events (participants affected / at risk) | 128/137 | 127/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=137) | Alvimopan 12 mg (N=143)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 2 (2) | 0 (0)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 2 (2) | 0 (0) — Resulted in two deaths
Cardio-Respiratory Arrest (Cardiac disorders) | 1 (1) | 0 (0) — Resulted in one death
Myocardial Infarction (Cardiac disorders) | 2 (2) | 2 (2) — Resulted in one death
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Gastrointestinal Angiodysplasia Haemorrhagic (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Enterocutaneous Fistula (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enterovesical Fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 7 (7) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Device Malfunction (General disorders) | 0 (0) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Sudden Death (General disorders) | 0 (0) | 1 (1) — Resulted in one death
Hepatic Cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis Chronic Active (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abdominal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Abdominal Infection (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 2 (2)
Clostridial Infection (Infections and infestations) | 2 (2) | 1 (1)
Clostridium Difficile Colitis (Infections and infestations) | 1 (1) | 1 (1)
Fungal Oesophagitis (Infections and infestations) | 0 (0) | 1 (1)
Fungal Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Incision Site Infection (Infections and infestations) | 1 (1) | 1 (1)
Pelvic Abscess (Infections and infestations) | 2 (2) | 3 (3) — Resulted in one death
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Postoperative Wound Infection (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 4 (4)
Pyelonephritis Acute (Infections and infestations) | 0 (0) | 1 (1)
Retroperitoneal Abscess (Infections and infestations) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 3 (3) | 1 (1) — Resulted in one death
Septic Shock (Infections and infestations) | 0 (0) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 5 (5)
Urinary Tract Infection Enterococcal (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection Staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 2 (2) — Resulted in one death
Abdominal Wound Dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal Anastomotic Leak (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Gun Shot Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Resulted in one death
Incisional Hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative Fever (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Postoperative Ileus (Injury, poisoning and procedural complications) | 28 (29) | 7 (8)
Postoperative Wound Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural Hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urinary Anastomotic Leak (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Urinary Retention Postoperative (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Wound Dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Clostridium Test Positive (Investigations) | 1 (1) | 0 (0)
Culture Positive (Investigations) | 1 (1) | 0 (0)
Staphylococcus Test Positive (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 7 (7) | 3 (3)
Failure To Thrive (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Throat Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Resulted in one death
Cerebral Infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy Peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Completed Suicide (Psychiatric disorders) | 0 (0) | 1 (1) — Resulted in one death
Delirium (Psychiatric disorders) | 1 (1) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 3 (3) | 3 (3)
Urinoma (Renal and urinary disorders) | 1 (1) | 0 (0)
Pelvic Fluid Collection (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — Resulted in one death
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) — Resulted in one death
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Abdominal Cavity Drainage (Surgical and medical procedures) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 5 (5) | 1 (1) — Resulted in one death
Hypotension (Vascular disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=137) | Alvimopan 12 mg (N=143)
Hypokalaemia (Metabolism and nutrition disorders) | 40 (40) | 27 (27)
Anaemia (Blood and lymphatic system disorders) | 34 (34) | 27 (27)
Nausea (Gastrointestinal disorders) | 32 (32) | 15 (15)
Hypocalcaemia (Metabolism and nutrition disorders) | 24 (24) | 21 (21)
Insomnia (Psychiatric disorders) | 20 (20) | 19 (19)
Pyrexia (General disorders) | 20 (20) | 18 (18)
Constipation (Gastrointestinal disorders) | 19 (19) | 21 (21)
Urinary Tract Infection (Infections and infestations) | 18 (18) | 11 (11)
Diarrhoea (Gastrointestinal disorders) | 17 (17) | 13 (13)
Hypomagnesaemia (Metabolism and nutrition disorders) | 17 (17) | 19 (19)
Oedema Peripheral (General disorders) | 17 (17) | 9 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 17 (17) | 10 (10)
Tachycardia (Cardiac disorders) | 16 (16) | 13 (13)
Flatulence (Gastrointestinal disorders) | 14 (14) | 7 (7)
Hyperglycaemia (Metabolism and nutrition disorders) | 14 (14) | 15 (15)
Hypotension (Vascular disorders) | 13 (13) | 13 (13)
Hypophosphataemia (Metabolism and nutrition disorders) | 12 (12) | 12 (12)
Anaemia Postoperative (Injury, poisoning and procedural complications) | 11 (11) | 9 (9)
Back Pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 1 (1)
Vomiting (Gastrointestinal disorders) | 11 (11) | 4 (4)
Hypertension (Vascular disorders) | 10 (10) | 13 (13)
Abdominal Pain (Gastrointestinal disorders) | 9 (9) | 6 (6)
Anxiety (Psychiatric disorders) | 9 (9) | 12 (12)
Dyspepsia (Gastrointestinal disorders) | 9 (9) | 6 (6)
Leukocytosis (Blood and lymphatic system disorders) | 9 (9) | 2 (2)
Postoperative Ileus (Injury, poisoning and procedural complications) | 9 (9) | 4 (4)
Haemoglobin Decreased (Investigations) | 8 (8) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 8 (8) | 6 (6)
Malnutrition (Metabolism and nutrition disorders) | 8 (8) | 3 (3)
Renal Failure Acute (Renal and urinary disorders) | 8 (8) | 6 (6)
Sinus Tachycardia (Cardiac disorders) | 8 (8) | 3 (3)
Blood Creatinine Increased (Investigations) | 7 (7) | 4 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 7 (7) | 5 (5)
Troponin Increased (Investigations) | 7 (7) | 5 (5)
Urine Output Decreased (Investigations) | 7 (7) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No